CLINICAL TRIAL: NCT04732845
Title: Phase I Clinical Trial of Human AntiCD19 Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Lymphoid Malignancies (Non-Hodgkin Lymphoma, Acute Lymphoblastic Leukemia, Chronic Lymphocytic Leukemia)
Brief Title: Human AntiCD19 Chimeric Antigen Receptor T Cells for Relapsed or Refractory Lymphoid Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Benjamin Tomlinson (Other)
Responsible Party: Sponsor-Investigator, Benjamin Tomlinson, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE2419
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Non Hodgkin Lymphoma; Acute Lymphoblastic Leukemia; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - NHL/CLL (Experimental): Upon enrollment, peripheral blood mononuclear cells will be collected, and T-cell selection and manufacture of CAR-T cells will be done.
  Participants will receive 60 mg/Kg/IV Cyclophosphamide on day -6 and 25 mg/m^2 Fludarabine from day -5 to day -3.
  Participants with CD19+ lymphomas and chronic lymphocytic leukemia will be enrolled on this arm sequentially in a 3 + 3 design starting with infusion of CAR-T cells at dose level 1 (DL1) on day 0.
  The maximum tolerated dose (MTD) will be determined and then 6 additional participants will be enrolled at the MTD.
  Interventions: Biological: Fully human anti CD19 CAR-T Cell Dose; Drug: Fludarabine; Drug: Cyclophosphamide
- Group B - ALL (Experimental): Upon enrollment, peripheral blood mononuclear cells will be collected, and T-cell selection and manufacture of CAR-T cells will be done.
  Participants will receive 60 mg/Kg/IV Cyclophosphamide on day -6 and 25 mg/m^2 Fludarabine from day -5 to day -3.
  Participants with Acute Lymphoblastic Leukemia (and lymphoblastic lymphoma as a solid tumor equivalent) will be enrolled on this arm sequentially in a 3 + 3 design starting with infusion of CAR-T cells at DL1 on day 0 and 7.
  The maximum tolerated dose (MTD) will be determined and then 6 additional participants will be enrolled at the MTD.
  Interventions: Biological: Fully human anti CD19 CAR-T Cell Dose; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Fully human anti CD19 CAR-T Cell Dose — Level -1 (1 x 10^5 cells/kg) Level 1 [Starting Dose] (5 x 10^5 cells/kg) Level 2 (1 x 10^6 cells/kg) Level 3 (2 x 10^6 cells/kg)
  Infusion of CAR-T cells will occur over 5-30 minutes.
Drug: Fludarabine — 25 mg/m2 daily from day -5 to -3
  Other Names: Fludara
Drug: Cyclophosphamide — 60mg/Kg on day -6
  Other Names: Cytoxan; Endoxan; Neosar; Procytox; Revimmune; Cycloblastin

SUMMARY:
The purpose of this study is to determine if it is possible to treat relapsed or refractory lymphoid malignancies (Non-Hodgkin Lymphoma, Acute Lymphoblastic Leukemia, Chronic Lymphocytic Leukemia) with a new type of T cell-based immunotherapy (therapy that uses the immune system to treat the cancer).

DETAILED DESCRIPTION:
This study seeks to determine the safety of the treatment of relapsed or refractory B cell lymphomas, relapsed/ refractory chronic lymphocytic leukemia and relapsed/refractory acute lymphoblastic leukemia with chimeric antigen receptor T cells targeting CD19 and to find the recommended phase II dose for this cellular therapy.

T cells are a type of white blood cell that helps the body fight infections. This treatment uses T cells already present within the body that have been modified outside of the body by a lentivirus and then returned to the participant by an infusion to target the cancer. Lentivirus is a family of viruses that can be used by scientists to alter cells, which then could be used to change the course of a disease. This type of treatment is sometimes referred to as adoptive cell transfer (ACT). In this study the specific type of cells that will be used is called human chimeric antigen receptor T cells (CAR-T cells). The CAR-T cells that will be reinfused to the body are modified using a lentivirus that is no longer active. The CAR-T cells will be returned to the body through an intravenous (IV) infusion. Another purpose of this study is to learn about the side effects and toxicities related to this treatment. Human CAR-T cell therapy is investigational (experimental) and works by removing T cells from the blood and modifying them to be able to target the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have relapsed or refractory non-Hodgkin lymphoma (NHL) (Group A - NHL/CLL), chronic lymphocytic leukemia (Group A - NHL/CLL) or acute lymphoblastic leukemia (Group B - ALL) treated with at least two lines of therapy. Disease must have either progressed after the last regimen or presented failure to achieve complete remission with the last regimen.
* The participant's malignancy is CD19 positive, either by immunohistochemistry or flow cytometry analysis on the last biopsy available or peripheral blood for circulating disease.
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
* Total bilirubin ≤ 1.5 times the institutional upper limit of normal unless bilirubin rise is due to Gilbert's syndrome (maximum 2 time normal) or of non-hepatic origin
* AST (SGOT) ≤ 3 times institutional upper limit of normal
* ALT (SGPT) ≤ 3 times institutional upper limit of normal
* Serum Creatinine ≤ 2 times the institutional upper limit of normal and creatinine clearance ≥ 30 mL/min (calculated or measured)
* Must have adequate pulmonary function as defined as pulse oximetry ≥ 92% on room air.
* Must have adequate cardiac function as defined as left ventricular ejection fraction≥ 40% in the most recent echocardiogram.
* Absolute Lymphocyte Count >100/microliter (uL)
* Participants (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 90 days after the human anti-CD19 CAR-T cell infusion. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the human anti-CD19 CAR-T cell infusion. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the human antiCD19 CAR-T cell infusion to avoid potential embryonal or fetal exposure. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods

Exclusion Criteria:

* Autologous transplant within 6 weeks of planned CAR-T cell infusion.
* Allogeneic stem cell transplant within 3 months of planned CAR-T cell infusion and patients must be off immunosuppressive agents.
* Active graft versus host disease.
* Active central nervous system or meningeal involvement by lymphoma or leukemia. Subjects with untreated brain metastases/central nervous system (CNS) disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Participants with a history of CNS or meningeal involvement must be in a documented remission by cerebrospinal fluid (CSF) evaluation and contrast-enhanced MRI imaging for at least 90 days prior to registration.
* Second active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast).
* A minimum of 28 days must have elapsed between prior treatment with investigational agent(s) and the day of lymphocyte collection.
* HIV seropositivity.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on screening bone marrow biopsy prior
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
* Participants with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
* History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2039-12-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of human anti-CD19 CAR-T cells | 24 months
  Recommended phase II dose of human anti-CD19 CAR-T cells

SECONDARY OUTCOMES:
Number of participants experiencing grade 3 or more adverse events | 18 months
  Toxicity profile for to infusion of fully human CAR-T cells, as measured by number of participants experiencing grade 3 or more adverse events
Number of participants experiencing dose limiting toxicities | 18 months
  Toxicity profile for to infusion of fully human CAR-T cells, as measured by number of participants experiencing dose limiting toxicities
Overall response rate (ORR) | 30 days after day 0 (first CAR-T treatment)
  ORR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Overall response rate (ORR) | 60 days after day 0 (first CAR-T treatment)
  ORR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Overall response rate (ORR) | 90 days after day 0 (first CAR-T treatment)
  ORR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Overall response rate (ORR) | 6 months after day 0 (first CAR-T treatment)
  ORR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Overall response rate (ORR) | 12 months after day 0 (first CAR-T treatment)
  ORR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Complete response rate (CR) | 30 days after day 0 (first CAR-T treatment)
  CR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Complete response rate (CR) | 60 days after day 0 (first CAR-T treatment)
  CR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Complete response rate (CR) | 90 days after day 0 (first CAR-T treatment)
  CR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Complete response rate (CR) | 6 months after day 0 (first CAR-T treatment)
  CR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Complete response rate (CR) | 12 months after day 0 (first CAR-T treatment)
  CR relapsed B cell malignancies treated with CAR-T cells targeting CD19
Progression Free Survival (PFS) | 30 days after day 0 (first CAR-T treatment)
  PFS from time of infusion
Progression Free Survival (PFS) | 60 days after day 0 (first CAR-T treatment)
  PFS from time of infusion
Progression Free Survival (PFS) | 90 days after day 0 (first CAR-T treatment)
  PFS from time of infusion
Progression Free Survival (PFS) | 6 months after day 0 (first CAR-T treatment)
  PFS from time of infusion
Progression Free Survival (PFS) | 12 months after day 0 (first CAR-T treatment)
  PFS from time of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tomlinson, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie or influence the results observed from the study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Link to be provided at time of article publication